CLINICAL TRIAL: NCT02586064
Title: Interpersonal Therapy for Veterans With PTSD
Brief Title: Comparative Effectiveness of Two Treatments for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Georgetown University (Other); Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1783-R; I01RX001783 (NIH)
Record Dates: First submitted 2015-10-20; First posted 2015-10-26 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; Veterans; Psychotherapy; Randomized Controlled Trial; Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interpersonal Psychotherapy for PTSD (Experimental): Relationally-focused intervention addressing PTSD symptoms and relationship dysfunctions, 12 weekly sessions
  Interventions: Behavioral: Interpersonal Therapy for PTSD
- Prolonged Exposure (Active Comparator): Exposure based intervention including exposure to memories and avoided places and activities
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: Interpersonal Therapy for PTSD — Relationally focused treatment that focuses on relationship problems that may be caused or maintained by PTSD symptoms. Consists of 12 individual weekly sessions of 45 to 50 minutes. Includes psycho-education, assessing which relationships (or lack of) are causing problems for the Veteran, and addressing the problem areas identified through specific strategies (e.g. communication analysis, decision analysis, role play). Final 2 sessions focus on consolidating what has been learned, what issues remain, identifying types of relationship triggers that could reactivate symptoms, and addressing feelings about termination.
  Arms: Interpersonal Psychotherapy for PTSD
Behavioral: Prolonged Exposure — Aim is to allow Veterans to re-experience traumatic events experienced during military service in a safe and supportive environment, and to re-engage in activities they have been avoiding. 12 individual weekly sessions of 90 minutes. Consists of psychoeducation, breathing retraining, imaginal exposure (repeated imaginal recall of the trauma including sensory details, and associated thoughts and feelings experienced during the trauma), and with trauma, and in vivo exposure (systematically confronting feared and avoided places and activities).
  Arms: Prolonged Exposure

SUMMARY:
Interpersonal problems such as relationship conflict and social isolation are common among Veterans with PTSD and serve as barriers to successful posttraumatic adjustment. The main interventions for PTSD at VA facilities, i.e., Prolonged Exposure, Cognitive Processing Therapy, and Trauma-Focused CBT, do not directly target these relationship difficulties and many Veterans do not complete these treatments. Couple and family approaches for PTSD address relationship problems, but logistical problems make it difficult for couples to attend sessions and these approaches do not involve Veterans who are socially isolated or unmarried. There is accumulating evidence that Interpersonal Psychotherapy (IPT) for PTSD may be effective in reducing symptoms and improving interpersonal functioning. This study, a randomized controlled trial, aims to provide evidence regarding whether IPT for PTSD could be a useful addition to current treatments delivered at the VA.

DETAILED DESCRIPTION:
The strong relationship between posttraumatic stress disorder (PTSD) and interpersonal problems is well documented. PTSD is highly associated with relationship discord, increased intimate partner violence, and difficulties in connecting with others, leading to social isolation. These types of conflicts, as well as the social withdrawal that is common among Veterans with PTSD, diminish the Veteran's opportunities for interaction with supportive others, and serve as a barrier to successful posttraumatic adjustment. Treatments that have been "rolled out" nationally in VAMCs, e.g., Prolonged Exposure, Cognitive Processing Therapy, and Trauma-Focused CBT, do not directly target these relationship difficulties. Furthermore, data show that only a limited number of Veterans has fully engaged with these interventions. Evidence-based interventions of couples therapy are available, but are not logistically feasible for many couples and do not address the problems of those who are socially isolated. This application proposes a randomized clinical trial of Interpersonal Psychotherapy (IPT-PTSD) as a treatment for Veterans with PTSD and relationship problems. Pilot data suggest that this type of treatment may provide a useful alternative strategy for Veterans who would prefer an individual, relationship-focused approach. The investigators propose comparing IPT-PTSD with Prolonged Exposure (PE), an evidence based treatment for PTSD used in the VHA system. The investigators hypothesize that IPT-PTSD will be statistically equivalent to PE in reducing PTSD symptom severity, and superior to PE in improving interpersonal functioning. IPT-PTSD is also hypothesized to be more effective than PE in improving social adjustment and quality of life. Exploratory analyses will examine whether IPT-PTSD is more effective than PE in reducing suicidal ideation, and will examine hypothesized mediators of improvement in PTSD symptoms in IPT-PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 18 or older
* Experienced trauma while deployed to a war zone
* Meet DSM-5 criteria for PTSD and a minimum CAPS-5 score of 23
* Have at least one area of relationship dysfunction
* Consent to be randomized

Exclusion Criteria:

* Current severe substance use disorder
* Current psychotic symptoms
* Current mania or un-medicated Bipolar Disorder
* Imminent threat of suicide or homicide
* Victim or perpetrator of severe domestic violence in the past 12 months
* Currently receiving Cognitive Behavioral Therapy for PTSD
* Psychotropic medication start or dosage change within the prior 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracie M. Shea, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
not developed yet
Supporting Information: Study Protocol
Time Frame: Following publication of primary and secondary study findings
Access Criteria: uncertain at this point

RESULTS

PARTICIPANT FLOW:
Groups:
- IPT-PTSD: Relationally-focused intervention addressing PTSD symptoms and relationship dysfunctions, 12 weekly sessions
  Interpersonal Therapy for PTSD: Relationally focused treatment that focuses on relationship problems that may be caused or maintained by PTSD symptoms. Consists of 12 individual weekly sessions of 45 to 50 minutes. Includes psycho-education, assessing which relationships (or lack of) are causing problems for the Veteran, and addressing the problem areas identified through specific strategies (e.g. communication analysis, decision analysis, role play). Final 2 sessions focus on consolidating what has been learned, what issues remain, identifying types of relationship triggers that could reactivate symptoms, and addressing feelings about termination.
Period: Overall Study
Arm/Group | IPT-PTSD | Prolonged Exposure
Started | 61 | 54
Completed | 43 | 26
Not Completed | 18 | 28
Not completed — Other Obligations | 6 | 6
Not completed — Other | 3 | 7
Not completed — Never Started | 3 | 3
Not completed — Lost Interest | 1 | 4
Not completed — Miscellaneous Life Issues | 0 | 5
Not completed — Infrequent Attendance | 2 | 1
Not completed — Timed Out | 2 | 0
Not completed — AUD relapse | 0 | 2
Not completed — Legal Issue | 1 | 0

BASELINE CHARACTERISTICS:
Population: While a total of 115 participants were randomized to IPT-PTSD (n=61) and Prolonged Exposure (n=54), 6 participants dropped before starting treatment therefore treatment analysis is based on a sample of 109 (58 IPT-PTSD and 51 Prolonged Exposure) participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPT-PTSD | Prolonged Exposure | Total
Number analyzed (Participants) | 58 | 51 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16) | 52 (15) | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 55 | 48 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 31 | 70
  Black | 14 | 17 | 31
  Other | 5 | 3 | 8
Clinician Assessment of PTSD Symptoms Version 5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — The Clinician Assessment of PTSD Symptoms Version 5 (CAPS-5) is used to assess change in PTSD symptoms in the past month. Item scores can range from 0 to 4 with total scores ranging from 0 to 80. Higher scores reflect more severe symptomatology.
  units on a scale | 36.3 (7.2) | 34.8 (7.4) | 35.6 (7.3)
PTSD Checklist Military Version 5 (PCL-M-5) [Mean (Standard Deviation); unit: units on a scale] — PTSD Checklist Military Version 5 (PCL-M-5) is a 20-item self-report measure that assesses DSM-5 symptoms of PTSD and PTSD symptom severity on a 5-point scale among military personnel. The self-report rating scale is 0-4 for each symptom, from 0 indicating that the subject endorses the frequency of this symptom as "Not at all" to 4 indicating the frequency as "Extremely." Scores can range from 0 - 80. Higher scores indicate more severe symptomatology. Population: Missing data from subjects at Baseline
  units on a scale
    number analyzed (Participants) | 57 | 49 | 106
    (all) | 48.0 (13.1) | 45.8 (12.7) | 47.6 (12.9)
Inventory of Interpersonal Functioning (IIP-32) [Mean (Standard Deviation); unit: units on a scale] — The Inventory of Interpersonal Functioning (IIP-32), is a 32 item questionnaire used to assess change in interpersonal functioning. Item scores range from 0 to 4 (0= Not at all to 4= extremely). Higher scores reflect worse interpersonal functioning.Total scores are based upon the mean of item ratings and range from 0 to 4.
  units on a scale | 1.53 (0.64) | 1.43 (0.56) | 1.48 (0.60)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire, the PHQ,-9, is a nine item version of the Primary Care Evaluation of Mental Health - MD Version (PRIME-MD) which contains the mood (PHQ-9) and anxiety modules in the original PRIME-MD. Scores can range from 0 "Not at all" to 3 "Nearly every day". Total scores range from 0 to 27 with higher scores indicating more severe depression.
  units on a scale | 15.2 (6.4) | 13.0 (7.3) | 14.2 (6.9)
Generalized Anxiety Disorder (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder - 7 Item (GAD-7) measures a participant's anxiety symptoms. Scores range from 0 to 3 with total score ranging from 0 - 21. Higher scores indicate more severe anxiety.
  units on a scale | 12.1 (5.8) | 11.6 (6.2) | 11.9 (6.0)
Multidimensional Scale of Perceived Social Support (MSPSS - Significant Other) [Mean (Standard Deviation); unit: units on a scale] — Multidimensional Scale of Perceived Social Support (MSPSS - Significant Other) is a 4 item subscale that measures perceived social support from the participant's significant other. Item scores range from 1 - 7 with total scores ranging from 4 - 28 with lower scores indicating lower perceived support.
  units on a scale | 4.9 (1.9) | 5.5 (1.2) | 5.2 (1.6)
Multidimensional Scale of Perceived Social Support (MSPSS) - Family [Mean (Standard Deviation); unit: units on a scale] — Multidimensional Scale of Perceived Social Support (MSPSS - Family) is a 4 item subscale that measures perceived social support from the participant's family. Item scores range from 1 - 7 with total scores ranging from 4 - 28 with lower scores indicating lower perceived support.
  units on a scale | 3.9 (1.8) | 4.6 (1.7) | 4.2 (1.8)
Multidimensional Scale of Perceived Support (MSPSS) - Friends [Mean (Standard Deviation); unit: units on a scale] — MSPPS - Friends is a 4 item subscale self report measure of perceived social support from friends scored on a scale from 1 - 7.that measures perceived social support from the participant's friends. Item scores range from 1 - 7 with total scores ranging from 4 - 28 with lower scores indicating lower perceived support.
  units on a scale | 3.9 (1.6) | 4.1 (1.5) | 4.0 (1.6)
Concise Health Risk Tracking (CHRT) Scale - Total [Mean (Standard Deviation); unit: units on a scale] — Concise Health Risk Tracking Scale (CHRT) Total is a 12-item self-report measure of suicidal ideation, hopelessness, and interpersonal attachment/social support. All items are rated on a 5-point scale (1 = strongly disagree, 5 = strongly agree).
  Scores range from a minimum value of 12 to a maximum value of 60 for our study. Higher scores indicate more risk for suicidal behavior.
  units on a scale | 27.6 (10.3) | 25.7 (10.4) | 26.8 (10.3)
Concise Health Risk Tracking (CHRT) - Propensity [Mean (Standard Deviation); unit: units on a scale] — Concise Health Risk Tracking Scale (CHRT) is a self-report measure of suicidal ideation, hopelessness, and interpersonal attachment/social support. All items are rated on a 5-point scale.
  The Propensity subscale score is the total of items 1 - 9 and can range for our study from a minimum value of 9 to a maximum value of 45. Higher scores indicate more risk for suicidal behavior.
  units on a scale | 22.8 (8.3) | 21.4 (8.8) | 22.1 (8.5)
Concise Health Risk Tracking (CHRT) - Suicidal Thoughts [Mean (Standard Deviation); unit: units on a scale] — Concise Health Risk Tracking Scale (CHRT) Suicidal Thoughts is a 12-item self-report measure of suicidal ideation, hopelessness, and interpersonal attachment/social support. All items are rated on a 5-point scale.
  The Suicidal Thoughts subscale score is the total of items 10 - 12 and can range for our study from a minimum value of 3 to a maximum value of 15. Higher scores indicate higher levels of suicidal behavior.
  units on a scale | 4.8 (2.6) | 4.3 (2.4) | 4.5 (2.5)
Work & Social Adjustment Scale (WSAS) Total [Mean (Standard Deviation); unit: units on a scale] — Work & Social Adjustment Scale (WSAS) Total is a self-report scale of functional impairment attributable to an identified problem in five different areas: ability to work, home management, social leisure, personal leisure, and maintaining close relationships.
  Scores range from a minimum value of 0 to a maximum value of 40, higher scores reflect more impairment in functioning.
  units on a scale | 24.0 (8.1) | 22.6 (9.6) | 22.8 (8.9)
WHO-QOL-BREF Item 1 Quality of Life [Mean (Standard Deviation); unit: units on a scale] — WHO Short Form Quality of Life Measure (WHOQOL-BREF) produces scores for four domains related to quality of life: physical health, psychological, social relationships and environment. Item scores range from 1 - 5. Higher scores reflect better quality of life.
  units on a scale | 3.1 (0.9) | 3.3 (1.0) | 3.2 (1.0)
WHO-QOL-BREF Item 2 Satisfaction with Health [Mean (Standard Deviation); unit: units on a scale] — WHO Short Form Quality of Life Measure (WHOQOL-BREF) produces scores for four domains related to quality of life: physical health, psychological, social relationships and environment. . Item scores range from 1 - 5. Higher scores reflect more satisfaction with health.
  units on a scale | 2.7 (1.0) | 2.8 (1.2) | 2.8 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale (CAPS-5)
Description: Structured interview for assessment of DSM-5 PTSD symptoms.
  Scores range from a minimum value of 0 to a maximum value of 80, higher scores mean a worse outcome.
Time Frame: Baseline, week 12 (end of treatment), 3 and 6 months posttreatment. End of Treatment assessment conducted following the last treatment session participant attended ideally after week 12 but could range from 9 to 20 weeks
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Difference Mean: Difference between mean of IPT-PTSD and Prolonged Exposure
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 36.3 (7.2) | 34.8 (7.4) | 1.52 (1.4)
  End of Treatment: number analyzed (Participants) | 50 | 32 | 82
  End of Treatment | 27.8 (9.8) | 28.2 (13.4) | -0.43 (2.57)
  Change: number analyzed (Participants) | 50 | 32 | 82
  Change | -8.1 (9.0) | -5.5 (11.3) | -2.56 (2.25)
  3 Month Post Treatment: number analyzed (Participants) | 42 | 32 | 74
  3 Month Post Treatment | 27.6 (12.4) | 26.3 (14.7) | 1.30 (3.16)
  6 Month Post Treatment | 25.6 (12.5) | 26.3 (14.3) | -0.61 (3.05)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.28, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; Test type: Equivalence — Confidence interval 95%, equivalence margin [-7,7]; Mean Difference (Final Values) = 1.52, Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.87, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD; Test type: Equivalence — Confidence interval 95%, equivalence margin [-7,7]; Mean Difference (Final Values) = -0.43, Standard Error of Mean 2.57
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Equivalence — Equivalence hypothesis was assessed using the confidence intervals for the mean differences compared to margins of equivalence (-7,7). The equivalence hypothesis was examined based on the difference between the amount of change from the baseline to the end of treatment on the CAPS between the two conditions. Confidence interval is -7.0 to 1.9; p = 0.26, t-test, 2 sided
Statistical Analysis 6: Comparison: IPT-PTSD vs Prolonged Exposure; Test type: Equivalence — Confidence interval 95%, equivalence margin [-7,7]; Mean Difference (Final Values) = -2.56, Standard Error of Mean 2.25
Statistical Analysis 7: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.68, t-test, 1 sided
Statistical Analysis 8: Comparison: IPT-PTSD vs Prolonged Exposure; Test type: Equivalence — Confidence interval 95%, equivalence margin [-7,7]; Mean Difference (Final Values) = 1.30, Standard Error of Mean 3.16
Statistical Analysis 9: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Follow Up; Test type: Other; p = 0.84, t-test, 1 sided
Statistical Analysis 10: Comparison: IPT-PTSD vs Prolonged Exposure; Test type: Equivalence — Confidence interval 95%, equivalence margin [-7,7]; Mean Difference (Final Values) = -0.61, Standard Error of Mean 3.05

2. Primary Outcome: Change in Inventory of Interpersonal Functioning (IIP-32)
Description: Self-report measure of Veterans' interpersonal difficulties.
  Scores range from a minimum value of 0 to a maximum value of 128, higher scores mean a worse outcome.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 3 and 6 months post-treatment. End of Treatment assessment conducted following the last treatment session participant attended ideally after week 12 but could range from 9 to 20 weeks
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
units on a scale
  Baseline | 1.53 (0.64) | 1.43 (0.56) | 0.11 (0.12)
  4 Week: number analyzed (Participants) | 48 | 35 | 83
  4 Week | 1.5 (0.5) | 1.4 (0.7) | 0.13 (0.14)
  8 Week: number analyzed (Participants) | 42 | 24 | 66
  8 Week | 1.3 (0.5) | 1.4 (0.7) | -0.12 (0.15)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 1.33 (0.63) | 1.21 (0.66) | 0.12 (0.14)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | -0.22 (0.57) | -0.15 (0.63) | -0.06 (0.13)
  3 Month Post Treatment: number analyzed (Participants) | 42 | 34 | 76
  3 Month Post Treatment | 1.2 (0.60) | 1.1 (0.60) | 0.17 (0.14)
  6 Month Post Treatment: number analyzed (Participants) | 43 | 35 | 78
  6 Month Post Treatment | 1.4 (0.60) | 1.1 (0.60) | 0.24 (0.14)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.36, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; 4-Week; Test type: Other; p = 0.34, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; 8-Week; Test type: Other; p = 0.43, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.09, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.41, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 6: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Superiority — Superiority hypotheses were assessed using the confidence interval for the mean differences (-0.33 to 0.20) compared to margin of superiority (-.05); p = 0.64, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5
Statistical Analysis 7: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.22, t-test, 1 sided; One sided 97.5% confidence interval, superiority margin was 0.5

3. Secondary Outcome: Change in PTSD Checklist for DSM-5 Military Version (PCL-M)
Description: Self report measure of DSM-5 PTSD symptoms.
  Scores range from a minimum value of 0 to a maximum value of 80, higher scores mean a worse outcome.
Time Frame: as for outcome 1
Population: Some participants skipped assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IPT-PTSD: Relationally-focused intervention addressing PTSD symptoms and relationship dysfunction.
- Difference Between Means: Difference between mean of IPT-PTSD and Prolonged Exposure
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 57 | 49 | 106
score on a scale
  Baseline | 48.0 (13.1) | 45.8 (12.7) | 2.15 (2.52)
  End of Treatment: number analyzed (Participants) | 47 | 34 | 81
  End of Treatment | 33.7 (15.9) | 35.5 (19.8) | -1.82 (3.96)
  Change: number analyzed (Participants) | 46 | 33 | 79
  Change | -12.8 (14.0) | -11.0 (18.8) | -1.75 (3.69)
  3-Month Follow Up: number analyzed (Participants) | 42 | 33 | 75
  3-Month Follow Up | 38.4 (17.4) | 36.2 (21.2) | 2.12 (4.46)
  6-Month Follow Up: number analyzed (Participants) | 42 | 33 | 75
  6-Month Follow Up | 36.1 (17.9) | 37.4 (20.0) | -1.35 (4.38)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.40, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.65, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.64, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.64, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.76, t-test, 1 sided

4. Secondary Outcome: Change in Patient Health Questionnaire (PHQ)
Description: Self report measure of mood and anxiety symptoms.
  Scores range from a minimum value of 0 to a maximum value of 27, higher scores mean a worse outcome.
Time Frame: as for outcome 2
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 15.2 (6.4) | 13.0 (7.3) | 2.15 (1.32)
  Week 4: number analyzed (Participants) | 48 | 32 | 80
  Week 4 | 13.9 (5.3) | 12.9 (7.2) | 1.0 (1.39)
  Week 8: number analyzed (Participants) | 41 | 24 | 65
  Week 8 | 11.1 (5.2) | 11.6 (6.9) | -0.50 (1.52)
  End of Treatment: number analyzed (Participants) | 48 | 34 | 82
  End of Treatment | 11.8 (6.5) | 10.3 (7.1) | 1.47 (1.51)
  Change: number analyzed (Participants) | 48 | 34 | 82
  Change | -3.1 (7.5) | -2.4 (7.0) | -0.74 (1.63)
  3 Month: number analyzed (Participants) | 41 | 33 | 74
  3 Month | 12.6 (5.7) | 10.3 (7.3) | 2.25 (1.51)
  6 Month: number analyzed (Participants) | 42 | 32 | 74
  6 Month | 13.2 (6.1) | 11.1 (7.2) | 2.09 (1.54)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.11, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; 4-Week; Test type: Other; p = 0.48, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; 8-Week; Test type: Other; p = 0.74, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.34, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.65, t-test, 1 sided
Statistical Analysis 6: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.14, t-test, 1 sided
Statistical Analysis 7: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.18, t-test, 1 sided

5. Secondary Outcome: Change in Multidimensional Scale of Perceived Social Support (MSPSS) - Significant Other
Description: Self-report measure of a participant's subjective social support with regards to a participant's significant other.
  For each subscale, the mean of items is reported therefore for the Significant Other Subscale: Sum across items 1, 2, 5, & 10, then divide by 4.Range can be from 1 - 7. Lower scores mean a worse outcome.
Time Frame: as for outcome 1
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 4.9 (1.9) | 5.5 (1.2) | -0.56 (0.31)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 4.9 (2.0) | 5.7 (1.5) | -0.74 (0.40)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | -0.13 (1.33) | -0.18 (0.99) | 0.05 (0.27)
  3 Month Post Tx: number analyzed (Participants) | 42 | 34 | 76
  3 Month Post Tx | 4.9 (1.7) | 6.0 (1.4) | -1.10 (0.36)
  6 Month Post Tx: number analyzed (Participants) | 43 | 35 | 78
  6 Month Post Tx | 5.2 (1.6) | 6.0 (1.3) | -0.76 (0.34)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.08, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.07, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.86, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.003, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.03, t-test, 1 sided

6. Secondary Outcome: Change in Multidimensional Scale of Perceived Social Support (MSPSS) - Family
Description: Self-report measure of a participant's subjective social support with regards to a participant's family.
  For each subscale, the mean of items is reported therefore for the Family Subscale: Sum across items 3, 4, 8, & 11 then divide by 4.Range can be from 1 - 7. Lower scores mean a worse outcome.
Time Frame: as for outcome 1
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 3.9 (1.8) | 4.6 (1.7) | -0.66 (0.33)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 4.4 (1.6) | 5.1 (1.7) | -0.75 (0.36)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | 0.34 (1.54) | 0.27 (1.76) | 0.07 (0.36)
  3 Month Post Tx: number analyzed (Participants) | 42 | 34 | 76
  3 Month Post Tx | 4.0 (1.7) | 5.5 (1.2) | -1.48 (0.34)
  6 Month Post Tx: number analyzed (Participants) | 43 | 35 | 78
  6 Month Post Tx | 4.5 (1.7) | 5.0 (1.8) | -0.56 (0.40)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.05, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.04, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.86, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p < 0.001, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.16, t-test, 1 sided

7. Secondary Outcome: Change in Multidimensional Scale of Perceived Social Support (MSPSS) - Friends
Description: Self-report measure of a participant's subjective social support with regards to a participant's family.
  For each subscale, the mean of items is reported therefore for the Friends Subscale: Sum across items 6, 7, 9, & 12 then divide by 4.Range can be from 1 - 7. Lower scores mean a worse outcome.
Time Frame: as for outcome 1
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 3.9 (1.6) | 4.1 (1.5) | -0.23 (0.30)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 4.4 (1.7) | 4.3 (1.8) | 0.14 (0.38)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | 0.5 (1.6) | 0.3 (1.8) | 0.20 (0.39)
  3 Month Post Tx: number analyzed (Participants) | 42 | 34 | 76
  3 Month Post Tx | 3.9 (1.5) | 4.4 (1.7) | -0.57 (0.37)
  6 Month Post Tx: number analyzed (Participants) | 43 | 35 | 78
  6 Month Post Tx | 4.3 (1.6) | 4.2 (1.8) | 0.10 (0.38)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.45, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.71, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.60, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.13, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.80, t-test, 1 sided

8. Secondary Outcome: Change in Concise Health Risk Tracking Scale - Total (CHRT)
Description: Self report measure of suicidal ideation and related symptoms.
  Our study used a response scale of 1 to 5. The CHRT has 12 items, and the total score has a possible range of 12 to 60. Higher scores indicate more suicidal ideation and risk.
Time Frame: as for outcome 1
Population: Some Veterans skipped assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 27.6 (10.3) | 25.7 (10.4) | 1.87 (1.98)
  End of Treatment: number analyzed (Participants) | 50 | 37 | 87
  End of Treatment | 25.4 (8.9) | 21.9 (10.9) | 3.49 (2.13)
  Change: number analyzed (Participants) | 50 | 37 | 87
  Change | -2.7 (8.9) | -3.5 (11.3) | 0.72 (2.16)
  3-Month Follow Up: number analyzed (Participants) | 42 | 34 | 76
  3-Month Follow Up | 27.1 (9.9) | 22.1 (9.8) | 5.04 (2.28)
  6-Month Follow Up: number analyzed (Participants) | 43 | 35 | 78
  6-Month Follow Up | 26.3 (9.7) | 23.5 (10.3) | 2.8 (2.27)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.35, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.11, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.74, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.03, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.22, t-test, 1 sided

9. Secondary Outcome: Change in Concise Health Risk Tracking Scale (CHRT) - Propensity
Description: The propensity subscale score includes 9 items assessing, hopelessness, self-worth and perceived social support, and the possible range for our study is 9 to 45
  Higher scores indicate worse outcome.
Time Frame: as for outcome 1
Population: Some Veterans skipped assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 22.8 (8.3) | 21.4 (8.8) | 1.40 (1.63)
  End of Treatment: number analyzed (Participants) | 50 | 37 | 87
  End of Treatment | 20.6 (7.6) | 17.9 (9.4) | 2.68 (1.82)
  Change: number analyzed (Participants) | 50 | 37 | 87
  Change | -2.6 (7.3) | -3.2 (9.3) | 0.64 (1.78)
  3-Month Follow Up: number analyzed (Participants) | 42 | 34 | 76
  3-Month Follow Up | 21.9 (7.9) | 18.0 (8.6) | 3.91 (1.89)
  6-Month Follow Up: number analyzed (Participants) | 43 | 35 | 78
  6-Month Follow Up | 21.4 (7.7) | 18.9 (8.8) | 2.46 (1.87)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.39, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.15, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.72, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.04, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.19, t-test, 1 sided

10. Secondary Outcome: Change in Concise Health Risk Tracking Scale (CHRT) - Suicidal Thoughts
Description: The CHRT Suicidal Thoughts subscale includes 3 items and has a possible range in our study from 3 to 15. Higher scores indicate higher suicidal thoughts.
Time Frame: as for outcome 1
Population: Some Veterans missed assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 4.8 (2.6) | 4.3 (2.4) | 0.47 (0.48)
  End of Treatment: number analyzed (Participants) | 50 | 37 | 87
  End of Treatment | 4.8 (2.4) | 4.0 (2.3) | 0.81 (0.50)
  Change: number analyzed (Participants) | 50 | 37 | 87
  Change | -0.16 (2.33) | -0.24 (2.83) | 0.08 (0.55)
  3-Month Follow Up: number analyzed (Participants) | 42 | 34 | 76
  3-Month Follow Up | 5.2 (2.9) | 4.1 (2.0) | 1.13 (0.57)
  6-Month Follow Up: number analyzed (Participants) | 43 | 35 | 78
  6-Month Follow Up | 4.9 (2.5) | 4.6 (2.5) | 0.33 (0.57)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.33, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.11, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.88, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.06, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.56, t-test, 1 sided

11. Secondary Outcome: Change in Work and Social Adjustment Scale (WSAS)
Description: Self report measure of functional impairment in five areas of functioning (work, home management, social leisure, personal leisure, close relationships.
  Scores range from a minimum value of 0 to a maximum value of 40, higher scores mean a worse outcome.
Time Frame: as for outcome 1
Population: Some Veterans missed completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Mean
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 24.0 (8.1) | 22.6 (9.6) | 2.40 (1.70)
  End of Treatment: number analyzed (Participants) | 50 | 37 | 87
  End of Treatment | 20.4 (10.8) | 15.8 (11.6) | 4.58 (2.41)
  Change: number analyzed (Participants) | 50 | 37 | 87
  Change | -3.5 (9.7) | -5.1 (9.9) | 1.58 (2.12)
  3 Month Post Tx: number analyzed (Participants) | 42 | 34 | 76
  3 Month Post Tx | 23.4 (9.2) | 15.5 (11.5) | 7.96 (2.37)
  6 Month Post Tx: number analyzed (Participants) | 43 | 35 | 78
  6 Month Post Tx | 23.4 (9.3) | 15.7 (11.6) | 7.73 (2.37)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.16, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.06, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.46, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Post Treatment; Test type: Other; p = 0.001, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.002, t-test, 1 sided

12. Secondary Outcome: Change in WHO Short Form Quality of Life Measure (WHOQOL-BREF) - Item 1 Quality of Life
Description: Measure of four domains related to quality of life: physical health, psychological, social relationships and environment. Data presented from Item 1 (Quality of Life)
  Scores range from a minimum value of 1 to a maximum value of 5, lower scores mean a worse outcome.
Time Frame: Difference between Baseline and End of Treatment means. End of Treatment assessment conducted following the last treatment session participant attended ideally after week 12 but could range from 9 to 20 weeks.
Population: Some Veterans missed completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 3.1 (0.9) | 3.3 (1.0) | -0.21 (0.18)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 73
  End of Treatment | 3.2 (0.9) | 3.2 (1.0) | 0.05 (0.20)
  Change: number analyzed (Participants) | 49 | 34 | 109
  Change | 0.04 (0.91) | -0.21 (0.98) | 0.25 (0.21)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.24, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.81, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.24, t-test, 1 sided

13. Secondary Outcome: Change in WHO Short Form Quality of Life Measure (WHOQOL-BREF) - Item 2 Satisfaction With Health
Description: Measure of four domains related to quality of life: physical health, psychological, social relationships and environment. Data presented from Item 2 (Satisfaction with Health).
  Scores range from a minimum value of 1 to a maximum value of 5, lower scores mean a worse outcome.
Time Frame: as for outcome 12
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 2.7 (1.0) | 2.8 (1.2) | -0.17 (0.21)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 2.6 (1.0) | 2.9 (1.1) | -0.29 (0.23)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | -0.12 (1.18) | 0.06 (1.23) | -0.18 (0.27)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.41, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.21, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.50, t-test, 1 sided

14. Secondary Outcome: GAD - 7 Generalized Anxiety Disorder
Description: Measure of generalized anxiety amongst participants over time.
  Scores range from a minimum value of 0 to a maximum value of 21, higher scores mean a worse outcome.
Time Frame: Baseline to 6 months posttreatment
Population: Some Veterans skipped completing assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPT-PTSD | Prolonged Exposure | Difference Between Means
Number analyzed (Participants) | 58 | 51 | 109
score on a scale
  Baseline | 12.1 (5.8) | 11.6 (6.2) | 0.44 (1.15)
  Week 4: number analyzed (Participants) | 47 | 34 | 81
  Week 4 | 12.2 (4.9) | 12.1 (5.5) | 0.06 (1.17)
  Week 8: number analyzed (Participants) | 42 | 22 | 64
  Week 8 | 9.6 (5.5) | 10.5 (6.4) | -0.84 (1.53)
  End of Treatment: number analyzed (Participants) | 49 | 34 | 83
  End of Treatment | 9.7 (5.7) | 9.0 (5.8) | 0.65 (1.29)
  Change: number analyzed (Participants) | 49 | 34 | 83
  Change | -2.3 (5.1) | -2.6 (6.3) | 0.25 (1.25)
  3 Month Follow Up: number analyzed (Participants) | 41 | 31 | 72
  3 Month Follow Up | 11.1 (6.0) | 9.6 (6.0) | 1.49 (1.43)
  6 Month Follow Up: number analyzed (Participants) | 41 | 34 | 75
  6 Month Follow Up | 11.0 (5.3) | 9.2 (5.6) | 1.80 (1.27)
Statistical Analysis 1: Comparison: IPT-PTSD vs Prolonged Exposure; Baseline; Test type: Other; p = 0.70, t-test, 1 sided
Statistical Analysis 2: Comparison: IPT-PTSD vs Prolonged Exposure; Week 4; Test type: Other; p = 0.96, t-test, 1 sided
Statistical Analysis 3: Comparison: IPT-PTSD vs Prolonged Exposure; Week 8; Test type: Other; p = 0.59, t-test, 1 sided
Statistical Analysis 4: Comparison: IPT-PTSD vs Prolonged Exposure; End of Treatment; Test type: Other; p = 0.61, t-test, 1 sided
Statistical Analysis 5: Comparison: IPT-PTSD vs Prolonged Exposure; Change; Test type: Other; p = 0.84, t-test, 1 sided
Statistical Analysis 6: Comparison: IPT-PTSD vs Prolonged Exposure; 3 Month Follow Up; Test type: Other; p = 0.30, t-test, 1 sided
Statistical Analysis 7: Comparison: IPT-PTSD vs Prolonged Exposure; 6 Month Post Treatment; Test type: Other; p = 0.16, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Baseline to 6 months post-treatment, an average of 9 months
Description: Definitions do not differ.
Arm/Group | IPT-PTSD | Prolonged Exposure
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/54
Serious Adverse Events (participants affected / at risk) | 8/61 | 3/54
Other Adverse Events (participants affected / at risk) | 0/61 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPT-PTSD (N=61) | Prolonged Exposure (N=54)
Inpatient Hospitalization - Alcohol (Psychiatric disorders) | 3 (3) | 2 (2)
Inpatient Hospitalization-Depression/Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Domestic Violence issue - Sustained minor injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Inpatient Hospitalization - Drugs (Psychiatric disorders) | 0 (0) | 1 (1)
Inpatient Hospitalization-Schizoaffective Disorder (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02586064/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02586064/ICF_001.pdf